CLINICAL TRIAL: NCT02563717
Title: A Randomised Controlled Trial of Delivery Room Intubation Rates Comparing a New System and T-piece Resuscitation System for Initial Stabilisation of Infants Born <28 Weeks
Brief Title: Comparison Of Respiratory Support After Delivery on Infants Born Before 28 Weeks Gestational Age
Acronym: CORSAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baldvin Jonsson (Other)
Responsible Party: Sponsor-Investigator, Baldvin Jonsson, Associate Professor and Clinical Director Karolinska University HospitalKarolinska University Hospital, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/927-31/4
Record Dates: First submitted 2015-09-24; First posted 2015-09-30 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Respiration; Insufficient or Poor, Newborn; Infant, Premature, Diseases
Keywords: Resuscitation; Positive-Pressure Respiration; Infant, Extremely Premature; Continuous Positive Airway Pressure; Intubation
MeSH Terms: conditions — Respiratory Aspiration; Infant, Premature, Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reference Device: T-piece System (Active Comparator)
  Interventions: Device: T-piece used for respiratory support (several manufacturers)
- Investigational Device: The New System (Active Comparator)
  Interventions: Device: New system used for respiratory support

INTERVENTIONS:
Device: T-piece used for respiratory support (several manufacturers) — Infants will receive support by a standard T-piece resuscitator system (manufacturer not dictated in protocol). Apart from the system used for respiratory support all patients will receive standard care (specified in management protocol)
  Other Names: Neopuff™ Infant T-Piece Resuscitator; T-piece Disposable Circuit Kit (GE Healthcare); Other T-piece manufacturers
  Arms: Reference Device: T-piece System
Device: New system used for respiratory support — Infants will receive support by the new system (manufactured by Inspiration Healthcare, UK). Apart from the system used for respiratory support all patients will receive standard care (specified in management protocol)
  Other Names: Manufacturing and CE-marking by Inspiration Healthcare, UK
  Arms: Investigational Device: The New System

SUMMARY:
Trial purpose: For infants born <28 weeks of age, can initial respiratory resuscitation with new system (low imposed work of breathing and prongs) reduce the frequency of delivery room intubations compared to standard treatment with T-piece resuscitator system (high imposed work of breathing and face mask)?

Trial summary: This is a randomised controlled trial of delivery room intubation rates comparing a new system and T-piece resuscitation system for initial stabilisation of infants born <28 weeks.

DETAILED DESCRIPTION:
The study is a two arm randomised comparison of two systems (T-piece device and the new system) for respiratory support after delivery of an infant born less than 28 weeks gestational age (GA). This multicentre trial will start at Karolinska University Hospital and other sites can join throughout the study period. The trial is academic with the coordinating investigator as sponsor. No company funding will be considered.

The new device has been designed for neonatal resuscitation and CE-marked for this intended use. The device is operated/handled in a similar way to existing devices and can provide support according to resuscitation guidelines.

During spontaneous breathing the continuous positive airway pressure (CPAP) provided with the new system is more pressure stable and has low imposed work of breathing. The benefits of decreased imposed work of breathing during resuscitation have not previously been investigated. The new system has the option of using prongs as the patient interface. Prongs have shown promising results in trials and have theoretical benefits. We hypothesis that the combined use of prongs and low imposed work of breathing could reduce the number of infants that need mechanical ventilation.

Screening for eligibility and consent will be performed on mothers with threatening delivery of an extremely premature infant (<28 weeks gestational age). There is no lower gestational age limit but patients should not be included if there is a decision to intubate prior to delivery or treatment limitations.

After a patient has been enrolled the randomisation will be on hold until delivery is imminent. Randomisation will be stratified on centre, gestational age and antenatal steroid treatment. The interventions cannot be blinded.

The management of respiratory support is according to international guidelines and a detailed description is provided in the clinical management appendix. The intervention is respiratory support for the first 10-30 minutes of life and will begin after birth when the infant is transferred to the resuscitation team. The intervention ends 1) when an infant is intubated (primary outcome), 2) after a minimum of 10 minutes support, with the randomized system, the patient is stable and breathing adequately, 3) at 30 minutes when the respiratory support can continue as decided by the clinicians (cross-over not allowed).

Apart from the system used for respiratory support all patients will receive standard care. No assessments or investigations of the trial subjects are planned. Data will be reported by the resuscitation team and collected from records.

The primary outcome is delivery room intubation or death. The secondary outcomes include time to intubation, use of surfactant, use of positive pressure ventilation, respiratory support at 72 hours and temperature on intensive care admission. Safety variables include pneumothorax, intraventricular haemorrhage and problems with ventilation and equipment.

All analysis will be on intention to treat and p<0.05 considered statistically significant. The primary outcome variable (delivery room intubation or death) will represent a 2x2 cross table and analysed with Pearson chi-square test. The secondary outcomes include Kaplan Meier analysis of time to intubation and comparisons of means for continuous variables. There are no predetermined subgroups. Subgroup analysis will be used to describe the population and to generate hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. Born <28 weeks gestational age at a university hospital
2. Delivery can be vaginal or with caesarean section and steroid prophylaxis to mother can be complete, incomplete or not given

Exclusion Criteria:

1. Decision on treatment limitations before randomisation
2. Decision to intubate infant made before delivery (for example local routine for infants born before 23 weeks GA)
3. Known airway, pulmonary, cardiac, gastro-intestinal tract malformations
4. Known neuromuscular disease
5. No study neonatologist available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Delivery room intubation or death | 0-30 minutes
  The primary outcome is delivery room intubation or death. Death has to be included in the primary outcome since patients that die may not always be intubated. The variable is a dichotomous outcome and reported by the resuscitation team.

SECONDARY OUTCOMES:
Time to primary outcome (intubation or death) | up to 72 hours of age
  The time (minutes:hours) that a patient reach primary outcome. Data reported by resuscitation team or collected at patient record review of the first three days of life. This is a safety endpoint.
Death | up to 72 hours of age
  The time (minutes:hours) that a patient died. Data reported by resuscitation team or collected at patient record review of the first three days of life. This is a safety endpoint.
Intra ventricular haemorrhage grade III or more | up to 72 hours of age
  The number of patients with an intra ventricular hemorrhage grade III or more. Data collected at patient record review of the first three days of life. This is a safety endpoint.
Airleaks and pneumothorax | up to 72 hours of age
  The number of patients with airleaks or pneumothorax during resuscitation or the first 72 hours of life. Data reported by resuscitation team or collected at patient record review of the first three days of life. This is a safety endpoint.
Failed ventilation | 0-30 minutes
  The number of patients with failed ventilation during resuscitation. Data reported by resuscitation team. This is a safety endpoint.
Device problems or malfunction | 0-30 minutes
  The instances that there was a problem with the randomized intervention. Data reported by resuscitation team. This is a safety endpoint. Device problems or malfunction activates the adverse events handling protocol.

OTHER OUTCOMES:
Surfactant use in delivery room (DR) and neonatal intensive care unit (NICU) | up to 72 hours of age
  The number of patients, method used and the number of doses that a patient received in the DR and NICU. Data reported by resuscitation team or collected at patient record review of the first three days of life.
The use of positive pressure ventilation (PPV) in delivery room | 0-30 minutes
  The number of patients that needed PPV during resuscitation. Data reported by resuscitation team.
Use of sustained inflation (not recommended) | 0-30 minutes
  The number of patients that were treated with a sustained inflation during resuscitation. This is not recommended and a violation of protocol. Data reported by resuscitation team.
Reason for DR intubation | 0-30 minutes
  The main reason for intubating patients in the DR during resuscitation. Data reported by resuscitation team.
Response to resuscitation measured by APGAR at 1, 5 and 10 minutes | 1-10 minutes
  The initial status of the patient and response to resuscitation measured by APGAR-scores (0-2 points on the five standard criteria). Data reported by resuscitation team.
Inspired oxygen level, oxygen saturation (SpO2) and level of CPAP support at 5 and 10 minutes | 5-10 minutes
  The initial status of the patient and response to resuscitation measured by need for oxygen (%), SpO2 (%) and the level of CPAP support (cm H2O). Data reported by resuscitation team.
Patient temperature on NICU admission | 10-180 minutes
  The temperature of the patients when they arrive to NICU (°C). Data collected at patient record review of the first three days of life.
Reason for NICU intubation | up to 72 hours of age
  The main reason for intubating patients in the NICU. Data collected at patient record review of the first three days of life.
Mechanical ventilation at any time <72 h | up to 72 hours of age
  The number of patients that has received mechanical ventilation at any time <72 hours. Data collected at patient record review of the first three days of life.
Mechanical ventilation or mode of non-invasive support at 72 h | at 72 hours of age
  The number of patients that had mechanical ventilation or non-invasive support at three days of age (including type of support). Data collected at patient record review of the first three days of life.
Decisions on treatment limitations during resuscitation | 0-30 minutes
  The number of patients that had any decision on limitations of treatment during resuscitation. Data reported by resuscitation team.
Withdrawal or withholding treatment | up to 72 hours of age
  The number of patients that had any decision on withdrawal or withholding treatment in the DR or NICU. Data collected at patient record review of the first three days of life.

CONTACTS AND LOCATIONS:
Overall Officials: Baldvin Jonsson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (6):
- Department of neonatology, University Hospital of Iceland, Reykjavik, Iceland
- Neonatal Unit, Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Stavanger University Hospital, Department of Pediatrics, Stavanger, Norway
- Department of Neonatology, Poznan University of Medical Sciences, Poznan, Poland
- Sweden (2):
  - University Hospital Linköping, Department of Pediatrics, Linköping
  - Karolinska University Hospital, Neonatology department, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared but method of sharing not decided

REFERENCES:
- [Derived] Donaldsson S, Palleri E, Jonsson B, Drevhammar T. Transition of Extremely Preterm Infants from Birth to Stable Breathing: A Secondary Analysis of the CORSAD Trial. Neonatology. 2023;120(2):250-256. doi: 10.1159/000528754. Epub 2023 Jan 23. PMID 36689927
- [Derived] Donaldsson S, Drevhammar T, Li Y, Bartocci M, Rettedal SI, Lundberg F, Odelberg-Johnson P, Szczapa T, Thordarson T, Pilypiene I, Thorkelsson T, Soderstrom L, Chijenas V, Jonsson B; CORSAD Trial Investigators. Comparison of Respiratory Support After Delivery in Infants Born Before 28 Weeks' Gestational Age: The CORSAD Randomized Clinical Trial. JAMA Pediatr. 2021 Sep 1;175(9):911-918. doi: 10.1001/jamapediatrics.2021.1497. PMID 34125148